CLINICAL TRIAL: NCT02507596
Title: Clinical and Radiographic Evaluation of Nano-crystalline Hydroxyapatite Silica Gel in the Treatment of Human Periodontal Intrabony Defects
Brief Title: Evaluation of Nano-crystalline Hydroxyapatite Silica Gel in Management of Periodontal Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of Oral Medicine and Periodontology, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nanobone_IBD
Record Dates: First submitted 2015-07-13; First posted 2015-07-24 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — NanoBone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nano-crystalline hydroxyapatite silica gel (Experimental): hydroxyapaptite bone graft with nano particle size in silica gel will be used to fill in the defect after opening a periodontal flap
  Interventions: Biological: Nano-crystalline hydroxyapatite silica gel
- Open flap debridement (Sham Comparator): an open periodontal flap without adding bone graft.
  Interventions: Procedure: open flap debridement

INTERVENTIONS:
Biological: Nano-crystalline hydroxyapatite silica gel — it is a type of synthetic bone graft.
  Other Names: Nanobone
  Arms: Nano-crystalline hydroxyapatite silica gel
Procedure: open flap debridement — a periodontal surgical procedure for the purpose of debridement.
  Other Names: OFD
  Arms: Open flap debridement

SUMMARY:
A clinical and radiographic evaluation of Nano-crystalline hydroxyapatite silica gel in comparison with open flap debridement for management of periodontal intrabony defects.

DETAILED DESCRIPTION:
Thirty patients suffering from advanced chronic periodontitis were included in this randomized controlled clinical trial. Each subject contributed matched two- or three-walled intrabony defects. Patients were equally assigned into the experimental group; Nano-crystalline hydroxyapatite silica gel or the negative control group;open flap debridement. Clinical and radiographic parameters were recorded at baseline and at 3 and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Severe chronic periodontitis patients.
* having at least one site with pocket depth ≥ 6 mm and clinical attachment level ≥ 5 mm, with radiographic evidence of bone loss as detected in periapical radiographs.

Exclusion Criteria:

* Pregnant women
* Subjects had <22 permanent teeth
* Having any given systemic disease
* Taking any type of medication and/or antibiotic therapy during the 3 months before the study
* Received periodontal treatment within the past 12 months Current or former smokers

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level | change from Baseline at 6 months
  Change from baseline in clinical attachment level in mm in chronic periodontitis patients at 6 month

SECONDARY OUTCOMES:
pocket depth | Baseline and 6 months
  Estimation of pocket depth in mm in chronic periodontitis patients at baseline and 6 months
bone defect area | Baseline and 6 months
  Estimation of bone fill defect area in mm square in chronic periodontitis patients at baseline and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Weam Battawy, MD, Study Chair — Lecturer of Oral Medicine and Periodontology; Noha Ghallab, MD, Principal Investigator — Associate Professor of Oral Medicine and Periodontology; Dalia AbdelHamid, MD, Study Director — Associate Professor of Biomaterials; Riham Hamdy, MD, Study Chair — Associate Professor of Oral and Maxillofacial Radiology
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Reynolds MA, Aichelmann-Reidy ME, Branch-Mays GL, Gunsolley JC. The efficacy of bone replacement grafts in the treatment of periodontal osseous defects. A systematic review. Ann Periodontol. 2003 Dec;8(1):227-65. doi: 10.1902/annals.2003.8.1.227. PMID 14971256
- [Background] Heinz B, Kasaj A, Teich M, Jepsen S. Clinical effects of nanocrystalline hydroxyapatite paste in the treatment of intrabony periodontal defects: a randomized controlled clinical study. Clin Oral Investig. 2010 Oct;14(5):525-31. doi: 10.1007/s00784-009-0325-x. Epub 2009 Aug 13. PMID 19680697
- [Background] Kasaj A, Rohrig B, Zafiropoulos GG, Willershausen B. Clinical evaluation of nanocrystalline hydroxyapatite paste in the treatment of human periodontal bony defects--a randomized controlled clinical trial: 6-month results. J Periodontol. 2008 Mar;79(3):394-400. doi: 10.1902/jop.2008.070378. PMID 18315420